CLINICAL TRIAL: NCT04836494
Title: A First-in-human, Randomized, Placebo-controlled, Single and Multiple Ascending Dose Escalation to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BBP-671 in Healthy Subjects and In Patients With Propionic Acidemia or Methylmalonic Acidemia
Brief Title: A First in Human, Dose Escalation Study to Evaluate the Safety and Tolerability of BBP-671 in Healthy Volunteers and Patients With Propionic Acidemia or Methylmalonic Acidemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: CoA Therapeutics, Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CoA-101
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers; Propionic Acidemia; Methylmalonic Acidemia; Organic Acidemia
MeSH Terms: conditions — Propionic Acidemia; Methylmalonic acidemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BBP-671 for SAD (Experimental): The SAD portion of the study will consist of up to 8 cohorts. Six (6) healthy male or female adult subjects will be randomized to receive BBP-671 per cohort (6:2 ratio, BBP-671:placebo).
  Interventions: Drug: BBP-671
- Placebo for SAD (Placebo Comparator): The SAD portion of the study will consist of up to 8 cohorts. Two (2) healthy male or female adult subjects will be randomized to receive matching placebo per cohort (6:2 ratio, BBP-671:placebo).
  Interventions: Drug: Placebo
- BBP-671 for MAD (Experimental): The MAD portion of the study will consist of up to 6 cohorts. Six (6) healthy male or female adult subjects will be randomized to receive BBP-671 per cohort (6:2 ratio, BBP-671:placebo).
  Interventions: Drug: BBP-671
- Placebo for MAD (Placebo Comparator): The MAD portion of the study will consist of up to 6 cohorts. Two (2) healthy male or female adult subjects will be randomized to receive matching placebo per cohort (6:2 ratio, BBP-671:placebo).
  Interventions: Drug: Placebo
- BBP-671 for SAD Food Effect (Experimental): Eight (8) healthy male or female adult subjects will be randomized to receive BBP-671.
  Interventions: Drug: BBP-671
- BBP-671 for PA and MMA Patients (Experimental): Up to sixteen (16) patients with either PA or MMA will receive BBP-671.
  Interventions: Drug: BBP-671

INTERVENTIONS:
Drug: BBP-671 — BBP-671, oral suspension
  Arms: BBP-671 for MAD; BBP-671 for SAD; BBP-671 for SAD Food Effect
Drug: Placebo — Placebo matching BBP-671
  Arms: Placebo for MAD; Placebo for SAD
Drug: BBP-671 — BBP-671, tablet
  Arms: BBP-671 for PA and MMA Patients

SUMMARY:
The purpose of this study is to assess the safety, tolerability, PK and PD of BBP-671 in healthy volunteers and patients with Propionic Acidemia or Methylmalonic Acidemia.

DETAILED DESCRIPTION:
This is the first-in-human study with BBP-671 and is designed to provide healthy subjects single- and multiple-dose and patient multidose safety, tolerability, PK, and PD data regarding BBP-671 for future clinical studies.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers):

* Subject is male or female 18 to 55 yrs old
* Subject has a BMI 18 to 32 kg/m^2
* Female and male subjects must use effective method of birth control
* Female subjects must have negative pregnancy test prior to first dose of study drug
* Subject must not have any clinically significant history or presence of ECG findings
* Subject must be in good general health

Inclusion Criteria (PA or MMA Patients):

* Patient is male or female 15 to 55 yrs old
* Patient has a BMI 18 to 32 kg/m^2
* Female and male patients must use effective method of birth control
* Female patients must have negative pregnancy test prior to first dose of study drug
* Patient must have confirmed PA or MMA diagnosis
* Patient with MMA must have elevated plasma MMA levels
* Patient is willing to provide access to medical records for the last 6-12 months of care prior to study initiation
* Patient is on consistent disease management and treatment regimen is stable for at least 30 days prior to study initiation.

Exclusion Criteria (Healthy Volunteers):

* Subject has used prescription drugs (contraceptive medications are allowed) within 4 weeks before first dose of study drug or over-the-counter medication within 7 days of the first dose of study drug
* Subject who is unable or unwilling to refrain from wearing contact lenses during participation in the study.
* Subject has a history of dry eye or eye surgery, including radial keratotomy and LASIK surgery.
* Subject who has taken the COVID-19 vaccine, the last vaccine dose must be at least 14 days prior to first dose of study drug.
* Subject has abnormal laboratory test results
* Subject has a baseline eGFR <90 mL/minute
* Subject has positive result for Hepatitis B, Hepatitis C, or HIV
* Female subject is non-pregnant and non-lactating
* Subject is a smoker or has used nicotine or nicotine-containing products
* Subject has a history of alcohol or drug abuse within 12 months prior to first dose of study drug and/or has a positive result prior to dosing or throughout the study
* Subject has donated blood or blood products >450mL within 30 days prior to study drug dosing
* Subject has a history of relevant drug or food allergies
* Subject has received study drug in another investigational study within 30 days of dosing
* Subject has undergone prior liver and/ or kidney transplant.

Exclusion Criteria (PA or MMA Patients):

* Patient has used prescription drugs (contraceptive medications are allowed) within 4 weeks before first dose of study drug or over-the-counter medication within 7 days of the first dose of study drug that is not part of their PA or MMA disease management and treatment
* Patient who has taken the COVID-19 vaccine, the last vaccine dose (or booster) must be at least 14 days prior to first dose of study drug.
* Patient is unable or unwilling to refrain from wearing contact lenses during participation in the study.
* Patient has a history of dry eye or eye surgery, including radial keratotomy and LASIK surgery.
* Patient has clinically significant abnormal laboratory test results unrelated to PA or MMA
* Patient has a baseline eGFR <60 mL/minute
* Patient has positive result for Hepatitis B, Hepatitis C, or HIV
* Female patient is non-pregnant and non-lactating
* Patient has a history of alcohol or drug abuse within 12 months prior to first dose of study drug and/or has a positive result prior to dosing or throughout the study
* Patient has donated blood or blood products >450mL within 30 days prior to study drug dosing
* Patient has a history of relevant drug or food allergies
* Patient has received study drug in another investigational study within 30 days of dosing
* PA patient has undergone prior liver and/ or kidney transplant. Prior liver and/or kidney transplant is allowed for patients with MMA.
* Patient has had a recent infection requiring system antibiotics within 4 weeks of Baseline or any active infection that precludes the patient from participation
* Patient has Grade 3 or 4 heart failure according to the Modified Ross Heart Failure Classification for Children or the New York Heart Association.
* Patient has been exposed to gene therapy for PA or MMA at any time prior to study entry.
* Patient is currently taking sensitive CYP3A4 substrates (e.g., tacrolimus or sirolimus)

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events following administration of BBP-671 | 49 days
BBP-671 concentration dependent change in change from baseline in QTcF | 49 days
Pharmacokinetic Assessments: Cmax | 49 days
  Time to maximum concentration (Cmax)
Pharmacokinetic Assessments: Tmax | 49 days
  Time to reach maximum observed plasma concentration (Tmax)
Pharmacokinetic Assessments: t1/2 | 49 days
  Plasma decay half-life (t1/2)
Pharmacokinetic Assessments: AUC0-tau | 49 days
  Area under the plasma concentration-time curve (AUC0-tau)
Pharmacokinetic Assessments: CL/F | 15 days
  Apparent clearance (CL/F)
Pharmacokinetic Assessments: Vz/F | 15 days
  Apparent volume of distribution (Vz/F)
Pharmacokinetic Assessments: CLr | 15 days
  Renal clearance (CLr)

SECONDARY OUTCOMES:
Food Effect: Cmax | 10 days
  Time to maximum concentration
Food Effect: Tmax | 10 days
  Time to reach maximum observed plasma concentration
Food Effect: AUC | 10 days
  Area under the plasma concentration-time curve
Pharmacodynamic Assessment: Whole blood, plasma, and urine biomarker concentrations will be quantified and summarized using appropriate descriptive parameters | 49 days
  Measurement will be done using liquid chromatography-tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Chair — VP Clinical Development, CoA Therapeutics, Inc., a Bridgebio company
Locations (3):
- United States (3):
  - Community Health Clinic, Topeka, Indiana
  - UPMC Children's Hospital of Pittsburg, Pittsburgh, Pennsylvania
  - PPD Development, LP, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Subramanian C, Frank MW, Sukhun R, Henry CE, Wade A, Harden ME, Rao S, Tangallapally R, Yun MK, White SW, Lee RE, Sinha U, Rock CO, Jackowski S. Pantothenate Kinase Activation Restores Brain Coenzyme A in a Mouse Model of Pantothenate Kinase-Associated Neurodegeneration. J Pharmacol Exp Ther. 2024 Jan 2;388(1):171-180. doi: 10.1124/jpet.123.001919. PMID 37875310